CLINICAL TRIAL: NCT04920669
Title: Can Dexmedetomidine Improve the Analgesic Duration and Efficacy of Erector Spinae Plane Block in Breast Cancer Surgeries?
Brief Title: Dexmedetomidine in Erector Spinae Block in Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Elsayed Hassan (Other)
Responsible Party: Sponsor-Investigator, Mohamed Elsayed Hassan, assistant professor of anesthesia and pain relief, National Cancer Institute, Egypt
Organization: National Cancer Institute, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AP2014-50103
Record Dates: First submitted 2021-05-30; First posted 2021-06-10 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain
Keywords: Erector spinae block.; dexmedetomidine.; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- erector spinae block (Experimental): erector spinae block with 20 ml bupivacaine
  Interventions: Procedure: erector spinae block with bupivacaine
- erector spinae block + dexmedetomidine (Experimental): erector spinae block with 19 ml bupivacaine + dexmedetomidine
  Interventions: Procedure: erector spinae block with bupivacaine + dexmedetomidine
- control group (No Intervention): standard general anesthesia without any block

INTERVENTIONS:
Procedure: erector spinae block with bupivacaine — Patients will receive a sonar-guided erector spinae plane block with 20 ml of bupivacaine 0.5%
  Arms: erector spinae block
Procedure: erector spinae block with bupivacaine + dexmedetomidine — Patients will receive a sonar-guided erector spinae plane block with 19 ml of bupivacaine 0.5%+ 1 ml dexmedetomidine
  Arms: erector spinae block + dexmedetomidine

SUMMARY:
60 female patients scheduled for breast cancer surgeries, allocated in 3 groups for erector spinae block with bupivacaine and erector spinae block with dexmedetomidine added to bupivacaine and control group. During anesthesia: total intraoperative fentanyl required will be recorded. After surgery the first time of request for analgesic will be recorded. after request of analgesia all patients will be connected to PCA device containing morphine solution, the amount of morphine consumed during the first 24 hours will be recorded.

DETAILED DESCRIPTION:
60 female patients scheduled for breast cancer surgeries, allocated in 3 groups for erector spinae block with bupivacaine and erector spinae block with dexmedetomidine added to bupivacaine and control group. During anesthesia: total intraoperative fentanyl required will be recorded. After surgery the first time of request for analgesic will be recorded. after request of analgesia all patients will be connected to PCA device containing morphine solution, the amount of morphine consumed during the first 24 hours will be recorded. Other secondary outcomes are numerical rating scales and incidence of opioid side effects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Female, aged (18-70) years
* Belongs to American Society of Anaesthesiologists physical status class II.
* Scheduled for breast cancer surgeries.

Exclusion Criteria:

* Patient refusal.
* Local infection at the site of the block.
* Cardiac dysfunction (ejection fraction <45%).
* Preexisting neurological or psychiatric disease, communication difficulties, inability to use the patient-controlled analgesia (PCA) device.
* Allergy to one of the study drugs.
* Pregnancy.
* Coagulopathy (PC <60% and platelet count<100.000).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Time to first request of analgesia | The first postoperative day
  Time from recovery of anesthesia till first request for analgesia to relive pain.

SECONDARY OUTCOMES:
Total morphine consumption in first postoperative 24 hours | First 24 postoperative hours
  The amount of morphine required to relieve pain will be recorded
Intraoperative fentanyl requirement | During anesthesia
  The amount of fentanyl required during anesthesia will be recorded
Numerical rating scale | The first 24 postoperative hours
  Numerical rating scale (from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain) will be recorded in different time intervals during the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Hassan, MD, Principal Investigator — National Cancer Institute, Cairo University, Egypt
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No